CLINICAL TRIAL: NCT03302754
Title: Precision Dosing of Alemtuzumab for Allogeneic Hematopoietic Cell Transplantation in Non-Malignant Diseases
Brief Title: Precision Dosing of Alemtuzumab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-2206
Record Dates: First submitted 2017-09-18; First posted 2017-10-05 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Allogeneic Hematopoietic Cell Transplantation
MeSH Terms: interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Alemtuzumab (Other): Patients less than 15kg will be given 0.6mg/kg alemtuzumab divided over days -14, -13, and -12 (0.2mg/kg/dose).
  Patients greater than 15kg will be given a 3mg "test" dose on day -14 in order to limit the first dose to no more than 3 mg per the manufacturer's recommendation. This will be followed by 0.23mg/kg/dose on days -13 and -12 (to equal a total dose of approximately 0.5-0.6mg/kg).
  Alemtuzumab will be drawn into a sterile syringe and given to patients subcutaneously.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Alemtuzumab (Campath®) is a recombinant DNA-derived humanized monoclonal antibody directed against CD52. Alemtuzumab is produced in mammalian cell (Chinese hamster ovary) suspension culture in a medium containing neomycin. Neomycin is not detectable in the final product. Alemtuzumab is a sterile, clear, colorless, isotonic pH 6.8-7.4 solution for injection. Alemtuzumab is supplied in single-use clear glass ampules containing 30 mg of Alemtuzumab in 3 mL of solution. Single use vial of alemtuzumab contains 30 mg alemtuzumab, 8 mg sodium chloride, 1.44 mg dibasic sodium phosphate, 0.2 mg potassium chloride, 0.2 mg monobasic potassium phosphate, 0.1 mg polysorbate 80, and 0.0187 mg disodium edetate dihydrate.
  Other Names: Campath

SUMMARY:
The purpose of this study is to conduct a pilot trial of a Precision Dosing approach to alemtuzumab dosing for allogeneic hematopoietic cell transplantation of patients with non-malignant diseases. The investigators will measure the ability to use a population PK model of alemtuzumab to target patient Day 0 alemtuzumab levels to 0.15-0.6ug/mL in a pilot study of 20 patients.

DETAILED DESCRIPTION:
The hypothesis is that the model-informed dosing regimen will prospectively allow the precision dosing of alemtuzumab to target Day 0 levels to fall between 0.15-0.6ug/mL in greater than 80% of patients. The investigators have chosen a conservative pilot study approach, and the aim is to achieve Day 0 alemtuzumab levels between 0.15-0.6ug/mL in greater than 60% of 20 patients enrolled in this pilot study based on a Simon two-stage design as detailed below.

A Simon two-stage design (Simon, 1989) is being used. The null hypothesis that 30% of patients will achieve a Day 0 alemtuzumab level between 0.15-0.6ug/mL will be tested against a one-sided alternative that the alemtuzumab dose modification will result in 60% of patients achieving a Day 0 alemtuzumab level between 0.15-0.6ug/mL. In the first stage, 7 patients will be accrued. If there are 2 or fewer patients that achieve Day 0 alemtuzumab levels within the range of 0.15-0.6ug/mL, the study will be stopped. Otherwise, 13 additional patients will be accrued for a total of 20. The null hypothesis will be rejected if 11 or more patients achieve a Day 0 level of 0.15-0.6ug/mL within the total 20 patients. This design yields a type I error rate of 0.04 and power of 0.82 when the true response rate is 0.60. The investigators will enroll up to 30 patients in order allow for subject withdrawal, but will stop enrollment once 20 patients reach Day 0.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are undergoing RIC HCT with alemtuzumab, fludarabine, and melphalan at CCHMC for treatment of a non-malignant disease.
2. Age ≥ 6 weeks to ≤ 30 years (at time of enrollment).
3. For the first 7 patients, patients must have a 10/10 HLA matched related or unrelated stem cell donor, or be receiving a CD34+ selected stem cell product. After the first 7 patients, any donor match may be allowed after data review by the PI and medical monitor.

Exclusion Criteria:

1. Patients with a history of anaphylaxis to alemtuzumab.
2. Patients who have previously received alemtuzumab and have not cleared alemtuzumab prior to the start of the preparative regimen.
3. Life expectancy less than 2 weeks.
4. Patients receiving dialysis.
5. Failure to sign informed consent and/or assent, or inability to undergo informed consent process.
6. It is not medically advisable to obtain the specimens necessary for this study.
7. Not able to tolerate subcutaneous dosing (patients with severe skin conditions such as epidermolysis bullosa).

Ages: 6 Weeks to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-03-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who have alemtuzumab levels in the optimal therapeutic range on Day 0. | 100 Days

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Marsh, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No